CLINICAL TRIAL: NCT00003847
Title: A Phase II Study of the Safety, Efficacy and Pharmacokinetics of VX-710 in Combination With Doxorubicin and Vincristine in Patients With Small Cell Lung Cancer (SCLC)
Brief Title: VX-710, Doxorubicin, and Vincristine for the Treatment of Patients With Recurrent Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067008; VX-98-710-006; DUMC-1450-98-9; NCI-V99-1537
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer; intermediate type small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — biricodar; Doxorubicin; Vincristine

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: biricodar dicitrate; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate

INTERVENTIONS:
Drug: biricodar dicitrate
Drug: doxorubicin hydrochloride
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy for the treatment of patients who have recurrent small cell lung cancer following treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Established the safety of VX-710 in combination with doxorubicin and vincristine for the treatment of patients with recurrent small cell lung cancer. II. Characterized the plasma pharmacokinetics of this regimen in patients. III. Established the ability of this regimen to improve the response rate to chemotherapy in patients who relapsed on front-line therapy. IV. Evaluated the multidrug resistance profile of these patients following this treatment regimen.

OUTLINE: This was a multicenter study. Stage I: Patients received VX-710 IV over 72 hours, followed by doxorubicin IV and vincristine IV four hours after initial VX-710. Vincristine was administered at half dose in the first 3-6 patients. If no more than 1 of 6 patients experienced a dose limiting toxicity in the half dose cohort, 3 additional patients received full dose vincristine. The maximum tolerated dose was defined as the dose preceding that at which 2 of 6 patients experienced a dose limiting toxicity. Stage II: Patients received VX-710 IV over 72 hours, followed by doxorubicin IV and full dose vincristine IV four hours after initial VX-710. Treatment continued for up to 6 courses every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients were followed every 3 months for up to 1 year.

PROJECTED ACCRUAL: A minimum of 35 and a maximum of 92 patients was to be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed oat cell or intermediate type small cell lung cancer Patients must have received prior therapy, with the following: Documented disease progression (new lesions or increased lesion size) after front line therapy No more than 1 prior chemotherapy regimen Complete or partial response to initial chemotherapy (must have lasted more than 60 days after end of therapy before relapse occurred) Bidimensionally measurable disease At least one lesion outside of irradiation field Pleural effusions are not measurable No brain or bone metastases as only measurable site No uncontrolled brain or other CNS metastases (surgical excision and/or radiotherapy)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: AST no greater than 2 times upper limit of normal Bilirubin no greater than 1.5 mg/dL Renal: Creatinine less than 1.3 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: Cardiac ejection fraction greater than 45% by MUGA or echocardiogram No uncontrolled ventricular arrhythmias Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No senile dementia or psychiatric disorders Not concurrent serious infection No major seizure disorder No grade 3 neuropathies No spinal cord compression No other concurrent unstable medical condition No other prior malignancies within past 5 years, except: Adequately treated basal or squamous cell skin cancer Any carcinoma in situ

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior doxorubicin or vincristine as first line treatment for small cell lung cancer Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to greater than 50% of bone marrow At least 30 days since prior radiotherapy Surgery: Not specified Other: No concurrent experimental drugs or anticancer therapies Concurrent medication for chronic medical conditions allowed (e.g., hypertension) No concurrent cimetidine, phenothiazines, phenobarbital, carbamazepine, troleandomycin, sulfinpyrazone, rifampin, Dilantin, and cyclosporine-A (or other P-gp inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1998-12; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Response Rate | Every 2 Cycles
  Analyzed via radiologic imaging according WHO criteria

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Harding, PhD, Study Chair — Vertex Pharmaceuticals Incorporated
Locations (9):
- United States (9):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Fallon Clinic Inc., Worcester, Massachusetts
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Gandhi L, Harding MW, Neubauer M, Langer CJ, Moore M, Ross HJ, Johnson BE, Lynch TJ. A phase II study of the safety and efficacy of the multidrug resistance inhibitor VX-710 combined with doxorubicin and vincristine in patients with recurrent small cell lung cancer. Cancer. 2007 Mar 1;109(5):924-32. doi: 10.1002/cncr.22492. PMID 17285598